CLINICAL TRIAL: NCT03356990
Title: Effects of Resistant Starch Diet on the Gut Microbiome in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 206708; 1P20GM121293 (NIH)
Record Dates: First submitted 2017-11-14; First posted 2017-11-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Resistant Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistant Starch (Experimental): Intervention:
  Dietary supplement will be taken every day for total of 2 weeks. Each participant will be take half the dose of Hi-Maze 260 or "High RS Gummy Chews" in the morning and the other half dose in the evening
  Adult participants are asked to introduce in their diet 30 grams of high RS supplement each day of the diet period (2 weeks).
  Children of age included between 5 and 9 years are asked to introduce in their diet 10 grams of high RS supplement each day of the diet period (2 weeks).
  Children of age included between 10 and 17 years are asked to introduce in their diet 15 grams of high RS supplement each day of the diet period (2 weeks).
  Interventions: Dietary Supplement: Resistant Starch

INTERVENTIONS:
Dietary Supplement: Resistant Starch — Dietary supplement will be taken every day for total of 2 weeks. Each participant will be take half the dose (one bag) of Hi-Maze 260 or "High RS Gummy Chews" in the morning and the other half dose (one bag) in the evening.

SUMMARY:
The investigators want to learn more about how to help people who have chronic kidney disease (CKD). This study will increase the investigators understanding of how diet affects factors that can slow the progression of kidney disease. The investigators are asking 30 adults and 30 children with stage 3 CKD to be part of this study. Participants will supplement their diet with resistant starch for two weeks. The investigators anticipate that the resistant starch will change the bacteria in the intestines to a more beneficial type of bacteria. The investigators will measure a product of these beneficial bacteria called butyrate. The investigators will also determine changes in the gut bacteria and products of the bacteria in the blood.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD), a progressive decline in kidney function, is a growing health problem: 13% of adults in the US have CKD. Among patients with CKD, the risk of progression to irreversible loss of kidney function (end-stage renal disease, ESRD) is about 1% per year. In addition, adjusted mortality is approximately four times greater among those with CKD compared to those without. For ESRD, apart from dialysis and kidney transplant, no treatment exists. CKD increases urea levels in bodily fluids leading to a dominance of urease-containing bacteria in the gut. Such dysbiosis results in decreased production of the short chain fatty acid, butyrate and decreased health of the colonic epithelial barrier. Consequently, bacterial toxins translocate into the bloodstream, promoting inflammation. Moreover, production of uremic toxins such as indoxyl and p-cresyl sulfates are also increased, resulting in further kidney injury.

CKD patients are prescribed a diet low in protein, fiber and symbiotic organisms, which reduces complications like hyperkalemia, but also contributes to the dysbiosis. Re-formulating the CKD diet may improve the clinical management of CKD. The investigators's overall hypothesis is that changes in the microbial diversity, xeno-proteins and xeno-metabolites correlate with CKD progression, and microbiome-directed therapies can be used to slow the disease. In this study, the investigators will determine the tolerability of supplemental resistant starch (RS). Secondary aims are to determine if a diet high in resistant starch changes fecal butyrate concentrations, the make-up of the gut microbiome and the concentrations in the blood of uremic toxins produced by the gut microbiome. This study will help in the design of a future study with the aim of understanding if a high resistant starch diet can slow the progression of chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult

  * Between the ages of 18 and 85 years old
  * Glomerular filtration rate estimated by creatinine clearance (eGFR Cr):between 59 and 30 ml/min for stage 3 CKD patients
  * Urine protein < 1 gram per day by 24-hour protein collection or urine protein-to-creatinine ratio <1 gram/gram or urine microalbumin to creatinine concentration less than 1000 mg/g.
* Children

  * Between the ages of 5 and 17 years
  * eGFR Cr between 30 and 59 (stage 3 CKD) using the revised Schwartz equation.
  * Urine protein < 1 gram per day by 24-hour protein collection or urine protein-to-creatinine ratio <1 gram/gram.

Exclusion Criteria:

Adult

* Age older than 85 years
* eGFR Cr > 59 ml/min or < 30 ml/min
* History of renal transplant
* Subject with diabetes (as defined by patient report, taking medications for the treatment of diabetes or as reported in the medical record)
* Use of antibiotics within 1 month
* Use of laxatives within 1 month
* Inflammatory bowel disease
* Irritable bowel syndrome
* Colorectal cancer
* Surgically removed bowel or presence of an ostomy
* Pregnancy
* Inability to obtain written informed consent
* Constipation
* Diarrhea

Children

* Age younger than 5 years
* eGFR > 59 ml/min and < 30 ml/min
* History of renal transplant
* Subject with diabetes (as defined by patient report, taking medications for the treatment of diabetes or as reported in the medical record)
* Use of antibiotics within 1 month
* Use of laxatives within 1 month
* Inflammatory bowel disease
* Surgically removed bowel or presence of an ostomy
* Pregnancy
* Constipation
* Diarrhea

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects that consume at least 90% of the dietary resistant starch (RS). | 2 weeks
  Packaging will be returned by the subject at the end of the time period in order to determine compliance.

CONTACTS AND LOCATIONS:
Overall Officials: John M Arthur, MD, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No